CLINICAL TRIAL: NCT05718466
Title: Prospective Study of Stereotactic Radiosurgery Using Diffusion-Weighted Abnormality Versus Chemotherapy for Recurrent/Progressive Glioblastoma After Second-line Chemotherapy
Brief Title: Stereotactic Radiology Versus Chemotherapy for Recurrent/Progressive Glioblastoma After Second-Line Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Salim Siddiqui, MD, PhD, Radiation Oncologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HFHS-C 11-01
Record Dates: First submitted 2014-02-26; First posted 2023-02-08 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Recurrent or Progressive Glioblastoma
Keywords: glioblastoma
MeSH Terms: conditions — Recurrence; Glioblastoma | interventions — Bevacizumab; Drug Therapy; Temozolomide; Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fractionated Radiosurgery and Bevacizumab (Experimental): FRS and Bev followed by Bev combined either Irinotecan or Temozolamide or Carboplatin or Etoposide until progression
  Interventions: Drug: Bevacizumab; Drug: Chemotherapy; Radiation: Fractionated radiosurgery
- Bev with Chemo (Active Comparator): Bev combined either Irinotecan or Temozolomide or Carboplatin or Etoposide until progression
  Interventions: Drug: Bevacizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Bevacizumab
Drug: Chemotherapy
  Other Names: Either irinotecan or temozolomide or carboplatin or etoposide
Radiation: Fractionated radiosurgery
  Arms: Fractionated Radiosurgery and Bevacizumab

SUMMARY:
This clinical trial is a prospective study of radiosurgery treatment for progressive GBM to test 1)the efficacy of radiosurgery for recurrent/progressive GBM compared to chemotherapy , and 2) the role of diffusion-weighted image (DWI) to predict the early tumor progression and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven intracranial glioblastoma multiforme with pathologic or imaging confirmation of tumor progression or regrowth after failure of two previous treatment regimens
* Initial low-grade glioma and a subsequent diagnosis of glioblastoma or gliosarcoma
* History and physical exam, including neurologic examination, within 4 weeks prior to registration

Exclusion Criteria:

• Warfarin or LMW heparin patients must have no active bleeding or pathological condition that carries a high risk of bleeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farzan Siddiqui, MD, Study Director — Henry Ford Hospital
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fractionated Radiosurgery and Bevacizumab: FRS and Bev followed by Bev combined either Irinotecan or Temozolamide or Carboplatin or Etoposide until progression
  Bevacizumab
  Chemotherapy
  Fractionated radiosurgery
- Bev With Chemo: Bev combined either Irinotecan or Temozolomide or Carboplatin or Etoposide until progression
  Bevacizumab
  Chemotherapy
Period: Overall Study
Arm/Group | Fractionated Radiosurgery and Bevacizumab | Bev With Chemo
Started | 18 | 17
Completed | 17 | 14
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fractionated Radiosurgery and Bevacizumab | Bev With Chemo | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (16.3) | 59.2 (8.3) | 55.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 14 | 11 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diagnosis [Count of Participants; unit: Participants]
  Anaplastic astrocytoma | 2 | 2 | 4
  Anaplastic oligodendroglioma | 0 | 2 | 2
  Glioblastoma | 16 | 13 | 29
Neoadjuvant RT Dose [Count of Participants; unit: Participants]
  54 | 0 | 1 | 1
  59.4 | 1 | 1 | 2
  60 | 17 | 15 | 32
Neoadjuvant Chemotherapy [Count of Participants; unit: Participants] | 16 | 17 | 33
On-Trial Chemotherapy [Count of Participants; unit: Participants]
  BEV+Carboplatin | 15 | 11 | 26
  BEV+etoposide | 1 | 0 | 1
  BEV+irinotecan | 0 | 0 | 0
  BEV+temozolomide | 1 | 2 | 3
  No trial chemotherapy | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Local Tumor Control
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fractionated Radiosurgery and Bevacizumab | Bev With Chemo
Number analyzed (Participants) | 17 | 15
Participants | 14 | 4

2. Primary Outcome: Overall Survival
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fractionated Radiosurgery and Bevacizumab | Bev With Chemo
Number analyzed (Participants) | 18 | 17
months | 7.2 [6.1 to 8.1] | 4.8 [1.7 to 7.6]
Statistical Analysis 1: Comparison: Fractionated Radiosurgery and Bevacizumab vs Bev With Chemo; Test type: Superiority; p = 0.11, Log Rank

3. Primary Outcome: Progression Free Survival
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fractionated Radiosurgery and Bevacizumab | Bev With Chemo
Number analyzed (Participants) | 18 | 17
months | 5.1 [4.1 to 6.2] | 1.8 [1.2 to 2.8]
Statistical Analysis 1: Comparison: Fractionated Radiosurgery and Bevacizumab vs Bev With Chemo; Test type: Superiority; p = 0.001, Log Rank

ADVERSE EVENTS:
Arm/Group | Fractionated Radiosurgery and Bevacizumab | Bev With Chemo
All-Cause Mortality (participants affected / at risk) | 15/18 | 14/17
Serious Adverse Events (participants affected / at risk) | 5/18 | 4/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fractionated Radiosurgery and Bevacizumab (N=18) | Bev With Chemo (N=17)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Grade 3
Headache (Nervous system disorders) | 1 | 0 — Grade 3
Nausea/Vomiting (General disorders) | 1 | 0 — Grade 3
New Onset Weakness (General disorders) | 1 | 0 — Grade 3
Seizure (Nervous system disorders) | 1 | 0 — Grade 3
Cerebral Edema (Nervous system disorders) | 0 | 1 — Grade 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 — Grade 3
Altered Mental Status (Nervous system disorders) | 0 | 1 — Grade 3
Intratumoral Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes